CLINICAL TRIAL: NCT00378170
Title: Laryngoscope Prototype Tested Against the Traditional Macintosh Blade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prototype vs Macintosh
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Anesthesia, Intravenous
Keywords: intubation; difficulty; Macintosh; dental damage; complications

INTERVENTIONS:
Device: intubation of patients undergoing elective surgery

SUMMARY:
The primary objective is to evaluate a knewly developed blade (for intubating patients about to undergo surgery) and compare it to the traditional Macintosh blade

DETAILED DESCRIPTION:
Intubation of patiens can be difficult, even impossible. It can result in different complications as damage to the teeth, lacerations of the mucosa, bleeding, fractures/luxations, hypoxia, hypercapnia, reflex bradycardia and in worst case braindamage and death.

The more difficult the intubation is the more frequent complicationrate. We believe to have developed a laryngoscopeblade that hopefully eases the intubationproces and thereby reduces the complicationrisk.

The patients included in this study is patients who are undergoing elective surgery requering intubation.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* ASA 1-III
* Patients undergoing elective surgery requering intubation at KAS Herlev

Exclusion Criteria:

* Prior difficult intubation indicating awake fiberoptic intubation
* pathology in the airways predicting difficult intubation
* columna cervicalis fractures
* pregnancy
* Requirement for Rapid sequence induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2006-01

PRIMARY OUTCOMES:
succes rate - immediate evaluation
difficulty - immediate evaluation

SECONDARY OUTCOMES:
Cormack & Lehane grading
Time to intubate
Interincissor gap
vissible complication

CONTACTS AND LOCATIONS:
Overall Officials: Ann Møller, consultant, Study Director
Locations (1):
- KAS Herlev university Hospital, Herlev, Herlev, Denmark